CLINICAL TRIAL: NCT06455722
Title: [68Ga]Ga-P15-041 PET/CT for Diagnosis and Prognostic Evaluation in Variety of Bone Tumors
Brief Title: [68Ga]Ga-P15-041 PET/CT in Variety of Bone Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-P15-041
Record Dates: First submitted 2023-12-10; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2023-12

CONDITIONS: Bone Tumor; Bone Metastases
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-P15-041; PET/CT (Experimental): Perform PET/CT after injecting [68Ga]Ga-P15-041
  Interventions: Drug: [68Ga]Ga-P15-041

INTERVENTIONS:
Drug: [68Ga]Ga-P15-041 — Intravenous injection of one dose of 111-148 MBq (3-4 mCi) [68Ga]Ga-P15-041. Tracer doses of [68Ga]Ga-P15-041 will be used to image lesions by PET/CT.
  Other Names: [68Ga]Ga-P15-041 PET/CT

SUMMARY:
Bone tumors refer to tumors that occur in the bone or its accessory tissues. Benign bone tumors usually reveal a good prognosis, while malignant bone tumors develop rapidly, have a poor prognosis and high mortality. Malignant bone tumors are also classified as primary tumor and secondary metastasis. Bone metastasis refers the metastasis of malignant tumors to the bone through lymph, blood or direct invasion to generate daughter tumors, which is the most common bone tumor. More than 40% of patients with malignant tumors will have bone metastasis, among which breast cancer, prostate cancer is more common. Early diagnosis of a various of bone tumors can lay the foundation for clinical implementation of effective treatment measures. The laboratory of Hank F. Kung at the University of Pennsylvania had developed a new generation of Gallium-68 labeled radiopharmaceutical P15-041 ([68Ga]Ga-P15-041) based on existing phosphonate-targeting molecular probes. Series of research results showed that [68Ga]Ga-P15-041 had high uptake in the bone cortex, blood and other tissues cleared quickly. Hence, [68Ga]Ga-P15-041 had the potential to become a new generation of excellent phosphonate molecular probes.

DETAILED DESCRIPTION:
Bone tumors refer to tumors that occur in the bone or its accessory tissues. Benign bone tumors usually reveal a good prognosis, while malignant bone tumors develop rapidly, have a poor prognosis and high mortality. Malignant bone tumors are also classified as primary tumor and secondary metastasis. Bone metastasis refers the metastasis of malignant tumors to the bone through lymph, blood or direct invasion to generate daughter tumors, which is the most common bone tumor. More than 40% of patients with malignant tumors will have bone metastasis, among which breast cancer, prostate cancer is more common. Early diagnosis of a various of bone tumors can lay the foundation for clinical implementation of effective treatment measures. The laboratory of Hank F. Kung at the University of Pennsylvania had developed a new generation of Gallium-68 labeled radiopharmaceutical P15-041 ([68Ga]Ga-P15-041) based on existing phosphonate-targeting molecular probes. Data from preclinical studies indicated that [68Ga]Ga-P15-041 shows additional advantages in rapid and easy complex formation compared to current agents. In preclinical experiments, [68Ga]Ga-P15-041 showed good bone resorption and rapid renal excretion in normal mice. Hong et al. prepared multiple clinical doses of [68Ga]Ga-P15-041 and successfully evaluated it in patients. Robert K. Doot et al. conducted dosemetric experiments on [68Ga]Ga-P15-041, and analyzed the radioactive distribution of the drug in normal organs and the dynamic change of the dose of the drug in the body over time. Series of research results showed that [68Ga]Ga-P15-041 had high uptake in the bone cortex, blood and other tissues cleared quickly. Hence, [68Ga]Ga-P15-041 had the potential to become a new generation of excellent phosphonate molecular probes.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed primary bone tumors or metastatic bone tumors
* signed written consent
* available other examinations such as bone scan or enhanced CT within 2 weeks

Exclusion Criteria:

* pregnancy
* breastfeeding
* known allergy against bisphosphonate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
detection capability | through study completion, an average of 6 months
  Record the number of bone tumor detected by [68Ga]Ga-P15-041 PET/CT, and compared it with other examinations such as bone scan and enhanced CT.
tumor uptake | through study completion, an average of 6 months
  Measure the standard uptake value of focal lesions on [68Ga]Ga-P15-041 PET/CT.

SECONDARY OUTCOMES:
survival | through study completion, an average of 6 months
  Follow up and record the time for patient's survival. To investigate the relationship between initial tumor uptake of focal lesions and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No